CLINICAL TRIAL: NCT06137911
Title: Safety, Tolerability and Pharmacokinetic Characteristics of JYP0061 in Healthy Adult Subjects After Single and Multiple Doses: a Single-center, Randomized, Double-blind, Placebo-controlled, Phase I Trial
Brief Title: Evaluation of Safety, Tolerability & Pharmacokinetics of JYP0061 in Healthy Adults.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou JOYO Pharma Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JYP0061M101
Record Dates: First submitted 2023-11-04; First posted 2023-11-18 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-04

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group A:JYP0061 15mg (Experimental): Experimental: JYP0061 Single ascending dose
  Interventions: Drug: JYP0061
- Group B:JYP0061 placebo comparator 15mg (Placebo Comparator): Placebo comparator: JYP0061 placebo comparator Single ascending dose
  Interventions: Drug: placebo
- Group C:JYP0061 food influence group 15mg (Experimental): Food influence group
  Interventions: Drug: JYP0061
- Group D:JYP0061 multiple ascending doses 30mg (Experimental): Multiple ascending doses
  Interventions: Drug: JYP0061
- Group E:JYP0061 placebo comparator food influence group 30mg (Placebo Comparator): Food influence group
  Interventions: Drug: placebo
- Group F:JYP0061 placebo comparator multiple ascending doses 30mg (Placebo Comparator): Multiple ascending doses
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: JYP0061 — JYP0061 orally administered
  Arms: Group A:JYP0061 15mg; Group C:JYP0061 food influence group 15mg; Group D:JYP0061 multiple ascending doses 30mg
Drug: placebo — Placebo orally administered
  Arms: Group B:JYP0061 placebo comparator 15mg; Group E:JYP0061 placebo comparator food influence group 30mg; Group F:JYP0061 placebo comparator multiple ascending doses 30mg

SUMMARY:
The goal of this clinical trial is to evaluate the safety, tolerability and pharmacokinetic characteristics of JYP0061 in healthy adult subjects. The main questions it aims to answer are: safety and tolerability of JYP0061 in healthy subjects, the pharmacokinetic characteristics after single and multiple doses and the effect of food on the pharmacokinetic characteristics. Participants will be treated with JYP0061 orally and safety and pharmacokinetic evaluations will be conducted according to the protocol.

DETAILED DESCRIPTION:
This study will be an double-blinded, single-center phase I clinical trial. After being informed about the study and potential risks, all subjects giving written informed consent will undergo a 2-week screening period to determine eligibility for study entry. And then subjects will be administered for single-dose treatment or 10-day multiple-dose treatment and 5-day safety follow up after the last dose of treatment. The safety and pharmacokinetic measures will be conducted according to the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years old (including both endpoints), healthy males or females;
* Male weight ≥50 kg, female weight ≥45 kg, body mass index (BMI) between 19-28kg/m^2 (including both endpoints);
* No significant abnormal clinical symptoms, normal physical examination, vital signs, 12-lead electrocardiogram (ECG), chest CT, ultrasound, and laboratory examination important indicators do not show clinically significant abnormalities;
* The participants (including partners) have no plans for childbearing from screening to 90 days after the last administration of the study drug, and are willing to take appropriate effective contraceptive measures (non-oral contraceptives);
* Fully understanding the study, voluntarily participate in the trial, and willingly sign the written informed consent.

Exclusion Criteria:

* Pregnant or lactating women;
* Individuals with special dietary requirements that cannot comply with a uniform diet;
* Suspected or confirmed allergy to any ingredients similar to the study drug or any ingredient in the study drug, or individuals with a history of allergic reactions;
* Past or current severe illness/abnormality (including but not limited to cardiac/cerebrovascular, respiratory, endocrine, metabolic, renal, hepatic, gastrointestinal, dermatological, malignant tumors, hematological, immune, rheumatological, neurological or psychiatric diseases), or any acute or chronic disease or physiological condition that could interfere with the trial results;
* Positive for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, Treponema pallidum antibody or human immunodeficiency virus (HIV) antibody; Participated in a clinical trial within the past 3 months;

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2021-09-26 (Actual); Primary Completion 2022-11-09 (Actual); Study Completion 2022-11-09 (Actual)

PRIMARY OUTCOMES:
The peak plasma concentration that JYP0061 achieves after dosing. | up to 4 weeks
  Evaluate patients' electrocardiogram data to detect whether the treatment causes maximum observed concentration of drug substance in plasma

SECONDARY OUTCOMES:
The time to reach the maximum concentration of JYP0061 in the bloodstream after administration. | up to 4 weeks
  Time when the maximum concentration is achieved

OTHER OUTCOMES:
The total drug exposure of JYP0061 from administration to an extrapolated infinite time, as represented by the area under the concentration-time curve. | up to 4 weeks
  Area under the concentration-time curve from time zero to infinity.in healthy subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Xuhui District Central Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No